CLINICAL TRIAL: NCT04376879
Title: Predicting the Need for Intubation in Hospitalised COVID-19 Patients (PRED ICU COVID19)
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A01076-33
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Step 1: creation of the score: Cohort for the creation of clinical-biological score to predict the risk of intubation in COVID-19
  Interventions: Other: Data monitoring for 48h within the first 24 hours of admission for COVID-19
- Step 2: validation of the score: Cohort for the validation of clinical-biological score to predict the risk of intubation in COVID-19
  Interventions: Other: Data monitoring for 48h within the first 24 hours of admission for COVID-19

INTERVENTIONS:
Other: Data monitoring for 48h within the first 24 hours of admission for COVID-19 — The admission variables and those constituting the predictive score (blood pressure, temperature, oxygenotherapy, biological analysis...) will be collected for 48 hours after enrolment (i.e within the first 24 hours of admission )

SUMMARY:
One of the main challenges of the health crisis caused by the COVID-19 epidemic is the availability of beds in intensive care units (ICUs) and, more importantly, the need for invasive mechanical ventilation (IVM) because the ICUs are currently reserved for intubated patients.

The experiences of both China and Italy indicate that a certain number of COVID-19 patients will require mechanical ventilation. However, the limited number of resuscitation beds and ventilators requires strict use of these scarce resources. As a significant proportion about 5% to 10%, of patients initially admitted to hospital with COVID-19 will require ventilation, it is essential to anticipate their need for resuscitation to improve the rare resource of beds and ventilator shortages in intensive care units.

The hypothesis of the study is that, in proven or suspected hospitalised and oxygen-requiring COVID-19 patients, an early predictive clinical score, calculated over the three first days of admission may allow for an earlier identification of patients who will require intubation and transfer to an intensive care unit for orotracheal intubation

ELIGIBILITY:
Inclusion Criteria:

* Proven or expected COVID-19 patients hospitalised in a non-intensive care unit for less than 24 hours,
* Patients requiring oxygen therapy,
* Age ≥ 18 years old.

Exclusion Criteria:

* Patients who are opposed to taking part in the study and who are opposed to the collection and use of the data that the study aims to collect.,
* Patients who can not be intubated for medical reasons,
* Pregnant women, parturient women or nursing mothers ,
* Adult person subject to a legal protection measure (guardianship, curatorship, judicial safeguard),
* Adults person who is unable to give consent and who is not subject to a legal protection measure,
* Persons deprived of their liberty by a judicial or administrative decision,
* Persons subject to psychiatric care under duress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Proven or expected COVID-19 patients hospitalised in a non-intensive care unit for less than 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2020-05-16 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
the number of intubations in COVID-19 patients initially hospitalised in wards | up to 1 month
  Primary outcome measure for the creation of the predictive score

SECONDARY OUTCOMES:
the number of intubations in COVID-19 patients initially hospitalised in wards. | up to 1 month
  Secondary endpoints for validation of the predictive score

CONTACTS AND LOCATIONS:
Overall Officials: Antoine KIMMOUN, MD-PhD, Study Chair — CHRU de NANCY; Jean Damien RICARD, MD-PhD, Study Chair — AP-HP, Louis Mourier Hospital; Julie JOSSE, PhD, Study Chair — Institut National de Recherche en Informatique et en Automatique; Patrick ROSSIGNOL, MD-PhD, Study Chair — CHRU de NANCY
Locations (2):
- France (2):
  - Louis Mourier hospital (AP-HP), Colombes
  - Brabois Hospital (CHRU de Nancy), Vandœuvre-lès-Nancy